CLINICAL TRIAL: NCT06808802
Title: A Phase 1, Open-label, Single-arm Study to Investigate the Effect of Retatrutide on Metoprolol Pharmacokinetics in Healthy Participants
Brief Title: To Investigate the Effect of Retatrutide (LY3437943) on Metoprolol Pharmacokinetics in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 27303; J1I-MC-GZQE (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-01-31; First posted 2025-02-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — retatrutide; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Retatrutide (Experimental): In period 1, participants will be administered a singe oral dose of metoprolol followed by a 1-week washout before retatrutide subcutaneous (SC) injection is given in period 2, followed by a second dose of metoprolol.
  Interventions: Drug: Retatrutide; Drug: Metoprolol

INTERVENTIONS:
Drug: Retatrutide — Administered subcutaneously (SC)
  Other Names: LY3437943
Drug: Metoprolol — Administered orally

SUMMARY:
The purpose of this study J1I-MC-GZQE is to measure the effect of retatrutide on the pharmacokinetics (PK) of metoprolol in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and vital signs
* Have a body mass index (BMI) within the range 22.0 to 35.0 kilogram per square meter (kg/m2) (inclusive) at screening

Exclusion Criteria:

* Have history of diabetes (except gestational diabetes) or current diagnosis of diabetes (any form), or have glycated hemoglobin (HbA1c) greater than or equal to (≥) 6.5% (48 millimole/mole (mmol/mol)
* Have a mean supine screening pulse rate of less than 45 or greater than 100 beats per minute (bpm) from 2 assessments. If a repeat measurement (mean of 2 assessments) shows values within the range of 45 to 100 bpm, the participant may be included in the trial
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, GI, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data
* Had any of the following cardiovascular conditions prior to screening: acute myocardial infarction, cerebrovascular accident, unstable angina, or hospitalization due to congestive heart failure

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under Concentration From Time Zero to Infinity (AUC[0-∞]) of Metoprolol | Day 1 to Day 3
  PK: AUC (0-∞) of Metoprolol
Pharmacokinetics (PK): AUC (0-∞) of Metoprolol with Retatrutide | Day 9 to Day 11
  PK: AUC (0-∞) of Metoprolol with Retatrutide
PK: Maximum Concentration (Cmax) of Metoprolol | Day 1 to Day 3
  PK: Cmax of Metoprolol
PK: Cmax of Metoprolol with Retatrutide | Day 9 to Day 11
  PK: Cmax of Metoprolol with Retatrutide

SECONDARY OUTCOMES:
Number of Participants with an Incidence of Treatment Emergent Adverse Events TEAEs (TEAEs) | Baseline to Day 44

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No